CLINICAL TRIAL: NCT01503645
Title: Epidemiology of Chinese Herb Nephropathy and Its Association With CYP2D6, CYP2C19, PXR, or MDR1 Polymorphism
Brief Title: Chinese Herb Nephropathy Epidemiology and Association With CYP2D6, CYP2C19, PXR, or MDR1 Polymorphism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 9461701139; 95D010
Record Dates: First submitted 2012-01-02; First posted 2012-01-04 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-01

CONDITIONS: Kidney Diseases
Keywords: kidney diseases; drugs, Chinese herbal; aristolochic acid; polymorphism, genetic
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Time Perspective: Cross-Sectional

SUMMARY:
1. Chinese herb nephropathy (CHN), a kind of kidney failure caused by Chinese herbs, may be related to the a component called aristolochic acid (AA).
2. AA may form AA-DNA adducts and accumulate in the kidney and ureter and cause kidney failure and/or cancer
3. Different enzymes have been reported to detoxify plant alkaloids or other components. Genes that regulate the production of these metabolic enzymes may affect the chance of CHN.
4. By comparing the differences in the polymorphisms of these genes between patient with CHN and control, we may find the changes that play a significant genetic factors for CHN.

ELIGIBILITY:
Inclusion Criteria:

* Patient with suspected Chinese herb nephropathy, and their family Control group match for sex age and geographic area (with or without herabla use)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People who use Chinese herb
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2006-05

CONTACTS AND LOCATIONS:
Overall Officials: Kwan-Dun Wu, MD, PhD, Study Chair — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - Far Estern Memorial Hospital, Banqiao District, Taipei
  - National Taiwan University Hospital, Taipei